CLINICAL TRIAL: NCT04029636
Title: Hyperpolarized 129Xe Magnetic Resonance Imaging for the Early Detection of Bronchiolitis Obliterans Syndrome (BOS) and Other Late Onset Non-infectious Pulmonary Complications (LONIPCs) Following Hematopoietic Stem Cell Transplantation
Brief Title: Hyperpolarized 129Xe MRI for the Assessment of BOS With Late Onset LONIPC
Acronym: BOS-MRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jane Turner, Principal Investigator, Hamilton Health Sciences Corporation
Other Study IDs: 5996
Record Dates: First submitted 2019-06-07; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Established LONIPC: The first cohort will comprise of patients with established LONIPCs and the investigative procedures in this study will provide data on the scope of abnormalities and pathology across the spectrum of these conditions.
  Interventions: Other: Inhaled Hyperpolarized Xenon-129
- Trajectory of LONIPC: The second, prospectively followed, cohort will provide data on the sequence and temporal development of these abnormalities, and therefore provide information on the trajectory of LONIPCs
  Interventions: Other: Inhaled Hyperpolarized Xenon-129

INTERVENTIONS:
Other: Inhaled Hyperpolarized Xenon-129 — How hyperpolarized 129Xe MRI measurements of lung structure and function change over time in a population at high risk for LONIPC related to their transplant

SUMMARY:
The development of bronchiolitis obliterans syndrome (BOS) and other late onset non-infectious pulmonary complications (LONIPCs) following hematopoietic stem cell transplantation (HSCT) is associated with a significantly worse prognosis, high disease burden, and excessive health resource utilization. In this proposal, the investigators plan to examine and compare different diagnostic modalities which can provide detailed physiological and anatomical characterization of LONIPCs.

DETAILED DESCRIPTION:
There is mounting evidence suggesting that current practice is failing to provide early detection of LONIPCs, before critical loss of lung function occurs. Furthermore, autopsy series in HSCT patients have revealed a wide spectrum of pulmonary pathology in different compartments of the lung (airway, parenchyma, interstitium) within the same individual. These findings imply that LONIPCs and the extent of their pulmonary involvement are under-recognized, which adversely impacts the clinical trajectory and outcomes of HSCT patients. These findings also suggest that the underlying pathophysiology is multi-faceted and diffuse, highlighting a need for a multi-modal approach to early detection, and better characterization of the spectrum of pulmonary involvement. In this study, we plan to examine and compare different diagnostic modalities which can provide detailed physiological and anatomical characterization of LONIPCs. We propose an observational study using hyperpolarized magnetic resonance imaging (MRI) to capture the anatomical and functional spectrum of LONIPCs post-HSCT. Hyperpolarized magnetic resonance imaging (MRI) is a novel and noninvasive functional imaging method, with the capacity to evaluate pulmonary structure and function. Inhaled hyperpolarized gas (129Xenon) maps focal areas of ventilation defects, a functional consequence of small airway obstruction, which often goes undetected on PFT in early disease states. It can provide additional information on alveolar structure and gas diffusion, lending insight into pathology in other compartments. Oscillometry technique (FOT) is a non-invasive technique using wave frequency to map out large and small airways, commonly used in pediatric pulmonology. We propose to examine the 2 novel modalities in HSCT patients with and without LONIPC/BOS. We hypothesize that the use of functional-structural imaging and FOT will provide better characterization and the extent of LONIPCs in early diseases states post-HSCT. These findings will provide invaluable insight into the pathophysiology of LONIPCs, providing a platform for future research into the early diagnosis and treatment of these high-burden diseases.

ELIGIBILITY:
Inclusion Criteria:

* For participants who have known LONIPC at enrollment (cross-sectional group):

  * Patient is 18 - 70 years old
  * Patient has received an allogenic HSCT
  * Diagnosed LONIPC

For participants who have no known LONIPC, but are at risk by virtue of recently-diagnosed cGVHD:

* Patient is 18 - 70 years old
* Patient has received an allogenic HSCT in the last 24 months
* Patient has a new diagnosis of cGVHD within the last 6 months by criteria of:

  * Moderate- or severe- cGVHD as per NIH consensus criteria, determined by a treating hematologist or
  * cGVHD requiring immunosuppression with prednisone at a dose of > 0.5mg/kg/day, or alternate steroid-sparing agent

Exclusion Criteria:

* For participants who have known LONIPC at enrollment (cross-sectional group):

  * Age less than 18 years or greater than 70 years of age
  * Current smoker (quit in the last 3 months)
  * Smoking history greater than 20 pack years
  * Presence of contraindications to pulmonary function testing including myocardial infarction within the last one month, hemoptysis, active communicable disease (e.g. TB), inability to follow commands, thoracic/abdominal/eye surgery within the last 3 months, pneumothorax, uncontrolled hypertension (SBP > 180, DBP > 110) or pulmonary embolism, other contraindication as determined by technical staff.
  * Pregnancy prior to or during study
  * In the opinion of the investigator, subject is mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
  * Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bio-prosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist/3T Manager)
  * In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia

For participants who have no known LONIPC, but are at risk by virtue of recently-diagnosed cGVHD:

* Age less than 18 years or greater than 70 years of age
* Known history of late onset non-infectious pulmonary complication (LONIPC) related to HSCT
* Current smoker (quit in the last 3 months)
* Smoking history greater than 20 pack years
* Presence of contraindications to pulmonary function testing including myocardial infarction within the last one month, hemoptysis, active communicable disease (e.g. TB), inability to follow commands, thoracic/abdominal/eye surgery within the last 3 months, pneumothorax, uncontrolled hypertension (SBP > 180, DBP > 110) or pulmonary embolism, other contraindication as determined by technical staff.
* Pregnancy prior to or during study
* In the opinion of the investigator, subject is mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bio-prosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist/3T Manager)
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. For participants who have known LONIPC at enrollment (cross-sectional group)
  2. For participants who have no known LONIPC, but are at risk by virtue of recently-diagnosed cGVHD
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The change detected in Ventilation Defect Percent (VDP) on 129Xe MRI imaging in cross-sectional and prospectively followed cohorts. | MRIs will be performed every three months for one year.
  129Xe Ventilation Defect Percent (VDP): For analysis of 129Xe static ventilation MR images we will employ the same approach as described by Kirby and colleagues to quantify the VDP to assess ventilation. VDP is expressed as a percentage.
The change detected in Apparent Diffusion Coefficients (ADC) on 129Xe MRI imaging in cross-sectional and prospectively followed cohorts. | MRIs will be performed every three months for one year.
  129Xe Apparent Diffusion Coefficients (ADC): For analysis of 129Xe diffusion-weighted MR images we will employ the same approach as described by Kirby and colleagues to quantify the ADC and generate ADC maps to assess airspace size. ADC is expressed in mm^2/s.
The change detected in Signal-to-noice Ration (SNR) on 129Xe MRI imaging in cross-sectional and prospectively followed cohorts. | MRIs will be performed every three months for one year.
  129Xe Signal-to-noise Ratio (SNR): The signal-to-noise ratio will be calculated as the mean signal intensity in a region of interest within the lung divided by the standard deviation in a region of interest outside of the lung.
The change detected in forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), total lung capacity (TLC), and residual volume (RV) in cross-sectional and prospectively followed cohorts. | Pulmonary Function Tests (PFTs) will be performed as clinically indicated, which in this study population will be every three months for two years.
  FVC, FEV1, TLC, and RV will be documented in litres (L) through pulmonary function testing.
The change detected in FEV1/FVC ratio and RV/TLC ratio in cross-sectional and prospectively followed cohorts. | PFTs will be performed as clinically indicated, which in this study population will be every three months for two years.
  FEV1/FVC ratio and RV/TLC ratio will be documented; these are ratios therefore and therefore do not have units.
The change detected in diffusion capacity of the lung for carbon monoxide (DLCO) and DLCO corrected for hemoglobin in cross-sectional and prospectively followed cohorts. | PFTs will be performed as clinically indicated, which in this study population will be every three months for two years.
  Diffusion capacity of the lung for carbon monoxide (DLCO) and DLCO corrected for hemoglobin will be recorded in L/min/mmHg.
The change detected in DLCO divided by alveolar volume (VA) [DLCO/VA, or transfer coefficient of the lung for carbon monoxide, KCO] in cross-sectional and prospectively followed cohorts. | PFTs will be performed as clinically indicated, which in this study population will be every three months for two years.
  DLCO divided by alveolar volume (DLCO/VA, or transfer coefficient of the lung for carbon monoxide [KCO]) will be recorded in mL/min/mmHg/L
The change detected in forced oscillometry technique (FOT) in cross-sectional and prospectively followed cohorts. | Oscillometry will be recorded every three months for one year.
  Results recorded in hertz (Hz)

SECONDARY OUTCOMES:
Change in airway resistance and reactance over time quantified by FOT | Oscillometry will be recorded every three months for one year.
  Measured in ohms (Ω)
Development of Bronchiolitis Obliterans Syndrome (BOS) | Development of BOS will be documented over the study's duration (2 years).
  The development of BOS will be defined using the National Institutes of Health (NIH) diagnostic criteria, and documented for all study participants (yes/no).
Development of clinical outcomes of death, hospitalization for respiratory cause, or respiratory failure. | Outcomes will be documented over the study's duration (2 years).
  The development of the above clinical outcomes will be documented for all study participants (yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien JW, Duncan S, Williams KM, Pavletic SZ. Bronchiolitis obliterans syndrome after allogeneic hematopoietic stem cell transplantation-an increasingly recognized manifestation of chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2010 Jan;16(1 Suppl):S106-14. doi: 10.1016/j.bbmt.2009.11.002. Epub 2009 Nov 5. PMID 19896545
- [Background] Walkup LL, Myers K, El-Bietar J, Nelson A, Willmering MM, Grimley M, Davies SM, Towe C, Woods JC. Xenon-129 MRI detects ventilation deficits in paediatric stem cell transplant patients unable to perform spirometry. Eur Respir J. 2019 May 2;53(5):1801779. doi: 10.1183/13993003.01779-2018. Print 2019 May. PMID 30846475
- [Background] Kirby M, Heydarian M, Svenningsen S, Wheatley A, McCormack DG, Etemad-Rezai R, Parraga G. Hyperpolarized 3He magnetic resonance functional imaging semiautomated segmentation. Acad Radiol. 2012 Feb;19(2):141-52. doi: 10.1016/j.acra.2011.10.007. Epub 2011 Nov 21. PMID 22104288
- [Background] Kirby M, Svenningsen S, Kanhere N, Owrangi A, Wheatley A, Coxson HO, Santyr GE, Paterson NA, McCormack DG, Parraga G. Pulmonary ventilation visualized using hyperpolarized helium-3 and xenon-129 magnetic resonance imaging: differences in COPD and relationship to emphysema. J Appl Physiol (1985). 2013 Mar 15;114(6):707-15. doi: 10.1152/japplphysiol.01206.2012. Epub 2012 Dec 13. PMID 23239874